CLINICAL TRIAL: NCT01638195
Title: A Feasibility Study: A Safety Evaluation of Renal Denervation Using Focused Therapeutic Ultrasound on Patients With Refractory Hypertension
Brief Title: A Safety Evaluation of Renal Denervation Using Focused Therapeutic Ultrasound on Patients With Refractory Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kona Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM11-002
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Externally Focused Ultrasound (Experimental)
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — Focused Ultrasound

SUMMARY:
This study is a prospective, single-institution trial wherein twenty subjects with refractory hypertension will receive the experimental focused ultrasound renal denervation therapy. Safety will be assessed by incidence and evaluation of serious adverse effects associated with the investigational procedure through 52-week evaluation of bilateral treatment. Clinical utility will also be evaluated by comparison pre and post therapy systolic and diastolic blood pressure and norepinephrine spillover.

DETAILED DESCRIPTION:
This study is a prospective, single-institution trial wherein each included subject will receive the experimental focused ultrasound renal denervation therapy. It will be conducted on a maximum of twenty adult male or female patients who meet the inclusion and exclusion criteria and have signed the informed consent form.

Safety is the primary endpoint of this study. Safety will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through the 52-week evaluation of bilateral treatment. Clinical utility is the secondary endpoint of this study. Clinical utility will be evaluated by assessing pre and post therapy systolic and diastolic blood pressure and norepinephrine (NE) spillover.

The study has been designed so that subjects are treated in a careful and stepwise fashion in order to minimize the potential risks associated with the investigational therapy. After completing baseline testing, the investigational focused ultrasound therapy will be unilaterally administered. Each subject is first treated on the right side. Renal angiograms are obtained after treatment is completed to ensure any resulting complications are quickly identified. After three weeks of treatment, the subject is further evaluated again with blood tests, EKG, angiogram and a norepinephrine spillover test. If any complications that preclude participation in the study are revealed, then additional treatment is halted. Upon safe treatment of the right renal artery, the left renal artery is then treated. Safety and functional evaluation occurs three weeks, and three and six months after completion of the last treatment. This sequential unilateral treatment scheme minimizes the potential risks to any given subject.

The second key factor in designing this study is the stepwise progression of applying the investigational therapy dose. Low dosing levels with established safety profile will first be applied before administering higher dosing levels. The low dosing level will be administered to the first ten subjects. The specified low dosing level was selected because it is just above the threshold value where renal denervation was detectable in the swine model, and patients participating in this cohort are expected to benefit from modest levels of renal neurolysis as measured by the norepinephrine spillover test. Only after five of the first ten subjects have been safely treated and evaluated at the 3-week follow-up evaluation may the remaining ten subjects (i.e., subjects #11 - 20) be treated with the higher dosing treatment. The specified higher dosing level was selected to induce increased renal neurolysis and thereby enable the expected escalated-dose response to be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject has systolic blood pressure of 160 mmHg or greater.
* Subject has refractory, stable hypertension despite being treated with at least three hypertensive drugs.
* Subject has two functioning kidneys, defined as eGFR ≥ 60 ml/min.

Exclusion Criteria:

* Subject has history of nephrectomy, kidney tumor or hydronephrosis.
* Subject has renal stenosis greater than 50%.
* Subject has presence of accessory renal artery with lumen ≥ 3 mm.
* Subject has a renal stent.
* Subject has end stage renal disease requiring dialysis or renal implant.
* Subject has Serum Cr > 3.0 mg/dL or equivalent calculated Glomerular Filtration Rate (GFR).
* Subject has a history of kidney stones.
* Subject has a history of abdominal surgery.
* Subject has a history of heterogeneities in the kidney such as cysts or tumors.
* Subject has a history of pyelonephritis.
* Subject has a history of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last six months.
* Subject has hemodynamically significant valvular heart disease.
* Subject has an implantable cardioverter defibrillator, pacemaker, neurostimulator or other device incompatible with MRI.
* Subject has a body weight > 150 kilograms.
* Subject has a target treatment depth > 14 cm.
* Subject is pregnant, nursing or intends to become pregnant during the trial period.
* Subject is currently enrolled in other potentially confounding research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety | 52 weeks post-treatment
  Safety will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through the 52-week evaluation of bilateral treatment. Included in this assessment will be the proportion of subjects with any of the following outcomes: (1) death, or (2) medical morbidity, including but not limited to renal artery aneurysm, stenosis, significant deterioration of renal function, fistulae or urethral stenosis.

SECONDARY OUTCOMES:
Blood Pressure Reduction | 52 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Whitbourn, M.D., Principal Investigator — St Vincent's Hospital
Locations (1):
- St. Vincent's Hospital, Melbourne, Victoria, Australia